CLINICAL TRIAL: NCT02821065
Title: TEC4Home: Telehealth for Emergency-Community Continuity of Care Connectivity Via Home-Telemonitoring
Brief Title: Telehealth for Emergency-Community Continuity of Care Connectivity Via Home-Telemonitoring
Acronym: TEC4Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kendall Ho, Lead, Digital Emergency Medicine; Professor, Department of Emergency Medicine, Faculty of Medicine, UBC, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H16-01076
Record Dates: First submitted 2016-05-24; First posted 2016-07-01 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single arm, pre-post study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Telemonitoring (Experimental): Patients will monitor their weight, blood pressure, oxygen saturation and symptoms with sensors and a tablet computer provided to them. Patients are asked to do this everyday for 60-days. A monitoring nurse receives and reviews the data electronically and will follow-up with the patient.
  Interventions: Device: Remote Patient Monitoring

INTERVENTIONS:
Device: Remote Patient Monitoring

SUMMARY:
Modern technology like computers, smartphones and the Internet enable patients to measure certain health indicators, like blood pressure and body weight, from the comfort of their own homes. This information can also be shared electronically with doctors and other healthcare providers to monitor remotely. This is called home health monitoring. In TEC4Home, we are developing a home monitoring solution for patients with heart failure to support their care and recovery at home after a visit to the emergency department. We hope to show that this solution decreases revisits to the emergency department and increases quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

PATIENT PARTICIPANTS:

* Have one or more typical symptoms of Heart Failure (i.e. dyspnoea at rest or minimal exertion (includes orthopnoea, reduced exercise tolerance)) AND
* Have one or more typical signs of Heart Failure (i.e. elevated jugular venous pressure, pulmonary crepitations, pleural effusions, peripheral oedema) AND
* Have one or more objective measures of heart failure:

Radiological congestion.

* Elevated BNP ≥ 400 pg/mL or NT-proBNP ≥ 1000 pg/mL.
* Reduced left ventricular ejection fraction <40% (or <45%) in previous 12 months.

Diastolic dysfunction including tissue Doppler E/e' ratio > 15 in previous 12 months.

* Pulmonary capillary wedge pressure >20 mmHg.
* Diuretic therapy. The additional value of diuretic therapy (IV or oral) is debatable, as presumably unlikely (or unsafe) that patient with genuine HF will be discharged without diuretic.

CLINICIAN PARTICIPANTS:

To be eligible to participate, clinician participants (i.e. ED physicians, family physicians and monitoring nurse(s)) must have referred or have a patient enrolled in the TEC4Home monitoring service.

Exclusion Criteria:

PATIENT PARTICIPANTS:

* Physical barriers e.g. unable to stand on scales.
* Cognitive impairment (e.g. MMSE <20), unless suitable caregiver support.
* Language (must be able to read and understand English), unless suitable caregiver support.
* Documented history of current and active substance misuse (within 3 months).
* Lack digital connectivity or landline phone connection.
* No regular care provider e.g. GP, or at least regular walk-in clinic.
* Existing intensive system of care: LVAD, transplant, dialysis.
* Anticipated improvement due to revascularization (PCI/CABG) or valve intervention during index hospitalization.
* Anticipated survival <90 days. Active palliative care, less-than level III care, disseminated malignancy.

CLINICIAN PARTICIPANTS:

Clinicians who do not have patients enrolled in the TEC4Home service or who themselves are not involved in the implementation or operation of the TEC4Home monitoring service will not be eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in number of emergency department revisits 90 day pre and 90 days post enrollment. | 90 days
  Hospital administrative data and self-reported data will be reviewed to assess the number of emergency department visits 90 day pre and 90 days post enrollment.
Change in the number of hospitalizations | 90 days
  Hospital administrative data and self-report data will be reviewed to assess the number of hospitalizations 90 day pre and 90 days post enrollment.
Change in the length of stay (in days) | 90 days
  Hospital administrative data and self-report data will be reviewed to assess the length of stay (measured in days) 90 day pre and 90 days post enrollment.
Mortality rate | 90 days
  The number of patients who pass away during the 90 day follow-up period will be recorded.

SECONDARY OUTCOMES:
Difference in quality of life (HF-specific) scores as assessed by the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ-12) scale | 90 days
  A 12 item disease-specific quality of life questionnaire will be administered to all participants for comparison pre-post enrollment.
Difference in quality of life (general) scores as assessed by the VR-12 | 90 Days
  A generic health-related quality of life questionnaire to be administered to all participants for comparison pre to post enrollment.
Difference in self-care efficacy scale scores as assessed by the European Heart Failure Self-care Behaviour Scale | 90 Days
  A 9 item scale to asses a patient's self-care behaviours and attitudes specific to Heart Failure will be administered to all participants for comparison pre-post enrollment.
Difference in costs and savings via administrative data and a self-report healthcare utilization survey. | 90 days
  Costs related to healthcare utilization and other health-related out of pocket and system costs will be assessed and compared 90 days pre to 90 days post enrollment
Impact of patient experience of care via surveys | 90 days
  Feedback from patients via survey questions to understand their experiences using the home health monitoring technology.
Impact of patient experience of care via interviews | 90 days
  Feedback from patients via interview questions to understand their experiences using the home health monitoring technology.
Impact on communication between healthcare providers and patients via surveys | 90 days
  Surveys about end-user experience will be used to collect feedback from patient participants, nurses, and other healthcare providers involved to understand the impact of home health monitoring on communication during the transition of care.
Impact on communication between healthcare providers and patients via interviews | 90 days
  Interviews about end-user experience will be used to collect feedback from patient participants, nurses, and other healthcare providers involved to understand the impact of home health monitoring on communication during the transition of care.

REFERENCES:
- [Derived] TEC4Home Healthcare Innovation Community. Supporting Heart Failure Patient Transitions From Acute to Community Care With Home Telemonitoring Technology: A Protocol for a Provincial Randomized Controlled Trial (TEC4Home). JMIR Res Protoc. 2016 Dec 18;5(4):e198. doi: 10.2196/resprot.5856. PMID 27977002